CLINICAL TRIAL: NCT06908785
Title: Utility of ROTEM® for Risk Stratification of Post-Invasive Procedure Hemorrhage in Patients With Cirrhosis (CIR-ROTEM)
Acronym: CIR-ROTEM
Status: Recruiting | Type: Observational
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Sponsor
Other Study IDs: CIR-ROTEM
Record Dates: First submitted 2025-03-25; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Cirrhosis, Liver
Keywords: Hemorrhage; Viscoelastic tests; Rotational thromboelastometry
MeSH Terms: conditions — Liver Cirrhosis; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EXPERIMENTAL GROUP: cirrhosis undergoing invasive procedures
  Interventions: Device: Rotational thromboelastometry

INTERVENTIONS:
Device: Rotational thromboelastometry — rotem

SUMMARY:
The assessment of post-procedural bleeding risk in cirrhosis remains a clinical challenge due to the lack of precise predictive tools and its high associated mortality. Although guidelines recommend a restrictive transfusion policy, adherence remains low, with a high rate of prophylactic transfusions despite unclear benefits. This multicenter, prospective, and observational study will evaluate the utility of ROTEM in bleeding risk stratification for cirrhotic patients with significant abnormalities in conventional hemostasis tests undergoing high-risk invasive procedures. The primary objective is to establish cut-off values with a high negative predictive value, optimizing transfusion decisions and reducing unnecessary blood product use. Additionally, the study will analyze the relationship between ROTEM, inflammation biomarkers, and coagulation factors, along with a cost-effectiveness analysis comparing different transfusion strategies. This will be the largest study to date assessing ROTEM in this setting, overcoming the limitations of previous studies, which have been mostly retrospective with heterogeneous populations and procedures. Its findings could contribute to the standardization of transfusion management in cirrhosis and improve healthcare resource efficiency. The widespread availability of ROTEM in other disciplines within the National Health System will facilitate its implementation in this clinical setting without requiring additional investment in equipment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 85 years.
* Clinical, analytical, elastographic, histological, and/or imaging criteria consistent with the diagnosis of hepatic cirrhosis.
* Undergoing a high-risk invasive procedure, either in an outpatient setting or during hospitalization.
* Platelet count below 50,000/μL or INR greater than 1.5 with a platelet count below 100,000/μL.
* Signature of informed consent.

Exclusion Criteria:

* Cirrhotic patients with acute-on-chronic liver failure (ACLF) as defined by EASL criteria, and patients admitted to Intensive Care Units. These patients are excluded because hemostatic alterations in ACLF and critically ill patients are different and more pronounced compared to those in outpatient or general medical ward settings.
* Chronic kidney disease stage ≥3.
* Presence and/or history of thromboembolic complications.
* Presence of non-hepatic tumors.
* Presence of any primary hematologic disease (including inherited coagulopathies or thrombophilia).
* Recent surgery (<8 weeks).
* History of organ transplantation, including liver transplantation.
* Pregnancy.
* Use of anticoagulants, antiplatelet agents other than acetylsalicylic acid, and/or antifibrinolytic therapy.
* Active disseminated intravascular coagulation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with cirrhosis undergoing invasive procedures
Sampling Method: Non-Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of post-procedural bleeding events within 28 days | 28 days after the procedure
  Number of participants with bleeding events occurring within 28 days after undergoing a high-risk invasive procedure. Bleeding will be classified according to the International Society on Thrombosis and Haemostasis (ISTH) criteria. ROTEM parameters (Clotting Time [CT], Clot Formation Time [CFT], Amplitude at 5/10 minutes [A5, A10], Maximum Clot Firmness [MCF], Maximum Lysis [ML], and Lysis Index at 30 minutes [LI30]) will be measured pre-procedure and analyzed to determine cut-off values with high negative predictive value for post-procedural bleeding.

CONTACTS AND LOCATIONS:
Locations (11):
- Spain (11):
  - Hospital universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital General Universitario Dr. Balmis de Alicante, Alicante
  - Hospital Clinic Barcelona, Barcelona
  - . Hospital de la Santa Creu i Sant, Barcelona
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Universitario de Cruces, Bilbao
  - Hospital Universitario de Burgos, Burgos
  - hospital Ramon y Cajal, Madrid
  - Hospital La Paz, Madrid
  - Huca, Oviedo
  - Hospital General Universitario de Toledo, Toledo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zanetto A, Rinder HM, Senzolo M, Simioni P, Garcia-Tsao G. Reduced Clot Stability by Thromboelastography as a Potential Indicator of Procedure-Related Bleeding in Decompensated Cirrhosis. Hepatol Commun. 2020 Dec 12;5(2):272-282. doi: 10.1002/hep4.1641. eCollection 2021 Feb. PMID 33553974
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines on prevention and management of bleeding and thrombosis in patients with cirrhosis. J Hepatol. 2022 May;76(5):1151-1184. doi: 10.1016/j.jhep.2021.09.003. Epub 2022 Mar 15. PMID 35300861
- [Background] Northup PG, Garcia-Pagan JC, Garcia-Tsao G, Intagliata NM, Superina RA, Roberts LN, Lisman T, Valla DC. Vascular Liver Disorders, Portal Vein Thrombosis, and Procedural Bleeding in Patients With Liver Disease: 2020 Practice Guidance by the American Association for the Study of Liver Diseases. Hepatology. 2021 Jan;73(1):366-413. doi: 10.1002/hep.31646. Epub 2021 Jan 20. No abstract available. PMID 33219529
- [Background] Northup PG, Friedman LS, Kamath PS. AGA Clinical Practice Update on Surgical Risk Assessment and Perioperative Management in Cirrhosis: Expert Review. Clin Gastroenterol Hepatol. 2019 Mar;17(4):595-606. doi: 10.1016/j.cgh.2018.09.043. Epub 2018 Sep 28. No abstract available. PMID 30273751
- [Background] Intagliata NM, Rahimi RS, Higuera-de-la-Tijera F, Simonetto DA, Farias AQ, Mazo DF, Boike JR, Stine JG, Serper M, Pereira G, Mattos AZ, Marciano S, Davis JPE, Benitez C, Chadha R, Mendez-Sanchez N, deLemos AS, Mohanty A, Dirchwolf M, Fortune BE, Northup PG, Patrie JT, Caldwell SH. Procedural-Related Bleeding in Hospitalized Patients With Liver Disease (PROC-BLeeD): An International, Prospective, Multicenter Observational Study. Gastroenterology. 2023 Sep;165(3):717-732. doi: 10.1053/j.gastro.2023.05.046. Epub 2023 Jun 2. PMID 37271290
- [Background] Pfisterer N, Schwarz M, Jachs M, Putre F, Ritt L, Mandorfer M, Madl C, Trauner M, Reiberger T. Endoscopic band ligation is safe despite low platelet count and high INR. Hepatol Int. 2023 Oct;17(5):1205-1214. doi: 10.1007/s12072-023-10515-y. Epub 2023 Apr 6. PMID 37024710
- [Background] Ronca V, Barabino M, Santambrogio R, Opocher E, Hodson J, Bertolini E, Birocchi S, Piccolo G, Battezzati P, Cattaneo M, Podda GM. Impact of Platelet Count on Perioperative Bleeding in Patients With Cirrhosis Undergoing Surgical Treatments of Liver Cancer. Hepatol Commun. 2022 Feb;6(2):423-434. doi: 10.1002/hep4.1806. Epub 2021 Oct 30. PMID 34716696
- [Background] Basili S, Raparelli V, Napoleone L, Talerico G, Corazza GR, Perticone F, Sacerdoti D, Andriulli A, Licata A, Pietrangelo A, Picardi A, Raimondo G, Violi F; PRO-LIVER Collaborators. Platelet Count Does Not Predict Bleeding in Cirrhotic Patients: Results from the PRO-LIVER Study. Am J Gastroenterol. 2018 Mar;113(3):368-375. doi: 10.1038/ajg.2017.457. Epub 2017 Dec 19. PMID 29257146
- [Background] Napolitano G, Iacobellis A, Merla A, Niro G, Valvano MR, Terracciano F, Siena D, Caruso M, Ippolito A, Mannuccio PM, Andriulli A. Bleeding after invasive procedures is rare and unpredicted by platelet counts in cirrhotic patients with thrombocytopenia. Eur J Intern Med. 2017 Mar;38:79-82. doi: 10.1016/j.ejim.2016.11.007. Epub 2016 Dec 15. PMID 27989373
- [Background] Bosch J, Thabut D, Albillos A, Carbonell N, Spicak J, Massard J, D'Amico G, Lebrec D, de Franchis R, Fabricius S, Cai Y, Bendtsen F; International Study Group on rFVIIa in UGI Hemorrhage. Recombinant factor VIIa for variceal bleeding in patients with advanced cirrhosis: A randomized, controlled trial. Hepatology. 2008 May;47(5):1604-14. doi: 10.1002/hep.22216. PMID 18393319
- [Background] Giannini EG, Greco A, Marenco S, Andorno E, Valente U, Savarino V. Incidence of bleeding following invasive procedures in patients with thrombocytopenia and advanced liver disease. Clin Gastroenterol Hepatol. 2010 Oct;8(10):899-902; quiz e109. doi: 10.1016/j.cgh.2010.06.018. Epub 2010 Jun 30. PMID 20601131
- [Background] Montalva E, Rodriguez-Peralvarez M, Blasi A, Bonanad S, Gavin O, Hierro L, Llado L, Llop E, Pozo-Laderas JC, Colmenero J; on behalf of the Spanish Society of Liver Transplantation and the Spanish Society of Thrombosis and Haemostasis. Consensus Statement on Hemostatic Management, Anticoagulation, and Antiplatelet Therapy in Liver Transplantation. Transplantation. 2022 Jun 1;106(6):1123-1131. doi: 10.1097/TP.0000000000004014. Epub 2022 Jan 4. PMID 34999660
- [Background] Under the auspices of the Italian Association for the Study of Liver Diseases (AISF) and the Italian Society of Internal Medicine (SIMI). Hemostatic balance in patients with liver cirrhosis: Report of a consensus conference. Dig Liver Dis. 2016 May;48(5):455-467. doi: 10.1016/j.dld.2016.02.008. Epub 2016 Feb 27. PMID 27012444
- [Background] Simonetto DA, Singal AK, Garcia-Tsao G, Caldwell SH, Ahn J, Kamath PS. ACG Clinical Guideline: Disorders of the Hepatic and Mesenteric Circulation. Am J Gastroenterol. 2020 Jan;115(1):18-40. doi: 10.14309/ajg.0000000000000486. PMID 31895720
- [Background] Patel IJ, Rahim S, Davidson JC, Hanks SE, Tam AL, Walker TG, Wilkins LR, Sarode R, Weinberg I. Society of Interventional Radiology Consensus Guidelines for the Periprocedural Management of Thrombotic and Bleeding Risk in Patients Undergoing Percutaneous Image-Guided Interventions-Part II: Recommendations: Endorsed by the Canadian Association for Interventional Radiology and the Cardiovascular and Interventional Radiological Society of Europe. J Vasc Interv Radiol. 2019 Aug;30(8):1168-1184.e1. doi: 10.1016/j.jvir.2019.04.017. Epub 2019 Jun 20. No abstract available. PMID 31229333
- [Background] Roberts LN, Lisman T, Stanworth S, Hernandez-Gea V, Magnusson M, Tripodi A, Thachil J. Periprocedural management of abnormal coagulation parameters and thrombocytopenia in patients with cirrhosis: Guidance from the SSC of the ISTH. J Thromb Haemost. 2022 Jan;20(1):39-47. doi: 10.1111/jth.15562. Epub 2021 Nov 8. PMID 34661370
- [Background] O'Shea RS, Davitkov P, Ko CW, Rajasekhar A, Su GL, Sultan S, Allen AM, Falck-Ytter Y. AGA Clinical Practice Guideline on the Management of Coagulation Disorders in Patients With Cirrhosis. Gastroenterology. 2021 Nov;161(5):1615-1627.e1. doi: 10.1053/j.gastro.2021.08.015. Epub 2021 Sep 25. No abstract available. PMID 34579936
- [Background] Riescher-Tuczkiewicz A, Caldwell SH, Kamath PS, Villa E, Rautou PE; Bleeding in liver diseases investigatorsdagger; Bleeding in liver diseases investigators. Expert opinion on bleeding risk from invasive procedures in cirrhosis. JHEP Rep. 2023 Dec 19;6(3):100986. doi: 10.1016/j.jhepr.2023.100986. eCollection 2024 Mar. PMID 38384669
- [Background] Desborough MJ, Hockley B, Sekhar M, Burroughs AK, Stanworth SJ, Jairath V; National Audit Collaborative. Patterns of blood component use in cirrhosis: a nationwide study. Liver Int. 2016 Apr;36(4):522-9. doi: 10.1111/liv.12999. Epub 2015 Nov 26. PMID 26537012
- [Background] Lu Y, Sun G, Liu X, Liu Z, Tan J, Hao Y, Shan G, Luo Q, Wang D, Xing Y, Zhang X, Gong J, Stanworth SJ, Wang J, Wen A. Plasma Transfusion in Patients With Cirrhosis in China: A Retrospective Multicenter Cohort Study. Transfus Med Rev. 2017 Apr;31(2):107-112. doi: 10.1016/j.tmrv.2016.11.006. Epub 2016 Dec 2. PMID 28063764
- [Background] Fortea JI, Puente A, Ezcurra I, Cuadrado A, Arias-Loste MT, Cabezas J, Llerena S, Iruzubieta P, Rodriguez-Lope C, Huelin P, Casafont F, Fabrega E, Crespo J. Management of haemostatic alterations and associated disorders in cirrhosis in Spain: A national survey. Dig Liver Dis. 2019 Jan;51(1):95-103. doi: 10.1016/j.dld.2018.06.003. Epub 2018 Jun 12. PMID 29960901
- [Background] Tosetti G, Farina E, Caccia R, Sorge A, Berzuini A, Valenti L, Prati D, Tripodi A, Lampertico P, Primignani M. Preprocedural prophylaxis with blood products in patients with cirrhosis: Results from a survey of the Italian Association for the Study of the Liver (AISF). Dig Liver Dis. 2022 Nov;54(11):1520-1526. doi: 10.1016/j.dld.2022.03.017. Epub 2022 Apr 23. PMID 35474168
- [Background] Malleeswaran S, Sivajothi S, Reddy MS. Viscoelastic Monitoring in Liver Transplantation. Liver Transpl. 2022 Jun;28(6):1090-1102. doi: 10.1002/lt.26352. Epub 2021 Dec 3. PMID 34724319